CLINICAL TRIAL: NCT05415124
Title: Presence or Absence of Blood in the GI Lumen - Correlating a HemoPill Acute Measurement With a Subsequent Endoscopic Finding
Brief Title: Presence or Absence of Blood in the GI Lumen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-00387
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Upper GI Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- HemoPill group (Experimental): Participants who have scheduled endoscopies will be given the HemoPill acute capsule and the HemoPill Receiver will be activated (connected to the HemPill). Approximately 20 to 60 minutes after HemoPill acute capsule ingestion, the endoscopy will start. The attending physician will proceed with the endoscopic intervention in accordance with clinical practice and NYU protocols, which is a standard procedure. In the case bleeding pathologies are found, these will be endoscopically treated as per clinical standard.For later evaluation of the HemoPill acute measurement, a statistical correlation of the obtained data from the HemoPill Acute measurement with the endoscopic findings will be performed. The HemoPill acute capsule travels through and leaves the body naturally
  Interventions: Device: HemoPill; Procedure: Endoscopy

INTERVENTIONS:
Device: HemoPill — The HemeoPill acute capsule is a small, single use, swallowable capsule with optical sensor. Blood detection by direct measurement of blood in the sensor gap, even in an unprepared digestive tract. Wireless transmission of measured values to the HemoPill Receiver. The maximum measuring time is 9 hours. The length of the capsule is 26.3 mm and the diameter is 7.0 mm.
Procedure: Endoscopy — Endoscopy is performed as scheduled.

SUMMARY:
Bleedings in the upper digestive tract are common. Usually, laboratory and clinical parameters are considered to establish a suspicion for a bleeding in the digestive tract and to estimate urgency of the situation. If these parameters suggest the presence of a bleeding in the digestive tract, endoscopies are often performed to further investigate a patient's status. The above-mentioned laboratory and clinical parameters are sometimes not specific enough to reliably identify a bleeding in the upper digestive tract. The HemoPill acute is capsule device, that has a built in sensor that detects blood in the upper digestive tract. This information is valuable for the medical personnel and complements the information that is obtained from other laboratory or clinical tests

DETAILED DESCRIPTION:
The purpose of the study was to access safety and accuracy of Hemopill and its receiver. Patients scheduled for endoscopy on the basis of suspected UGIB are generally eligible for inclusion into the trial. After patient screening, information and obtaining informed consent, a patient is enrolled into the trial. Shortly before the scheduled endoscopy is performed, the patient ingests a HemoPill acute. Endoscopy is performed as scheduled. Blood within the GI lumen is identified if present and pictures are taken. Pathologies, if found, are treated as per clinical standard. The HemoPill acute measurement regarding presence or absence of blood in the GI lumen is compared to observations made during endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled for endoscopy due to suspicion of UGIB based on clinical and / or laboratory findings
* Signed informed consent
* Age ≥ 18 years
* Willingness and ability to participate in the study procedure

Exclusion Criteria:

* Contraindications to the use of the HemoPill acute, such as:
* Known gastrointestinal obstruction, stricture, fistula, or diverticula
* Dysphagia or other swallowing disorders
* Pregnancy
* Incapacity to provide informed consent
* In patients with cardiac pacemakers and other implanted medical devices

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Debordeaux, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to Melissa.latorre@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HemoPill Group
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HemoPill Group
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (22.087)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With True Positive Results
Description: HemoPill acute measurement positive; Endoscopy measurement positive. HemoPill acute measurement indicates presence of blood; Endoscopy identifies fresh blood or hematin in the GI lumen
Time Frame: 1 hour after endoscopy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | HemoPill Group
Number analyzed (Participants) | 13
Participants | 3

2. Primary Outcome: Number of Participants With False Positive Results
Description: HemoPill acute measurement positive; Endoscopy measurement negative. HemoPill acute measurement indicates presence of blood; Endoscopy does not identify fresh blood or hematin in the GI lumen.
Time Frame: 1 hour after endoscopy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | HemoPill Group
Number analyzed (Participants) | 13
Participants | 3

3. Primary Outcome: Count of Participants With True Negative Results
Description: HemoPill acute measurement negative; Endoscopy measurement negative. HemoPill acute measurement does not indicate presence of blood; Endoscopy does not identify fresh blood or hematin in the GI lumen in quantities > 20 mL; Minimum latency of 20 minutes achieved.
Time Frame: 1 hour after endoscopy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | HemoPill Group
Number analyzed (Participants) | 13
Participants | 5

4. Primary Outcome: Count of Participants With False Negative Results
Description: HemoPill acute measurement negative; Endoscopy measurement positive. HemoPill acute measurement does not indicate presence of blood in the GI lumen; Endoscopy identifies fresh blood or hematin in the GI lumen in quantities > 20 mL; minimum latency of 20 minutes achieved.
Time Frame: 1 hour after endoscopy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | HemoPill Group
Number analyzed (Participants) | 13
Participants | 2

ADVERSE EVENTS:
Time Frame: Endoscopy procedure (Day 1)
Description: Adverse event information collected during endoscopy procedure.
Arm/Group | HemoPill Group
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT05415124/Prot_SAP_000.pdf